CLINICAL TRIAL: NCT04222569
Title: Determination of the Optimal Spontaneous Breathing Trial During Weaning of Mechanical Ventilation: a Randomized and Personalized Cross Over Physiologic Study in the Perioperative and Critically Ill Patient
Brief Title: Determination of the Optimal Spontaneous Breathing Trial During Weaning of Mechanical Ventilation
Acronym: GLOBAL WEAN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: sufficient number of patients to meet objectives
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RECHMPL19_0197
Record Dates: First submitted 2019-12-09; First posted 2020-01-10 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Intensive Care Unit; Invasive Mechanical Ventilation; Ready to Wean From Ventilation
Keywords: Intensive Care Unit; Critical Care; Mechanical Ventilation Weaning; Spontaneous Breath Trial; Rehabilitation

STUDY DESIGN:
Intervention Model Description: Each patient, serving as their own control, realize three SBT for 15 minutes: T-piece, PSV 7 cmH2O without PEEP and PSV 0 cmH2O without PEEP. The order is randomized. The randomization is stratified on pathology. For avoid a carry-over effect, a wash-out period of baseline ventilation for 10 minutes will be respected between trials. The humidification device is a heated humidifier, linked to the ventilator. Data are recorded before (guarantee of real return to baseline) and after each SBT.
  Then, extubation is decided by clinician in charge, in accordance with guidelines. A 30 min of resting period is respected before. Data are recorded before and 20 minutes after extubation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- T-piece and PSV 7 PEEP 0 and PSV 0 PEEP 0 (Experimental): First T-piece trial for 15 min. After 10 min of rest, PSV 7 cmH2O and PEEP 0 cmH2O trial for 15 min. After 10 min of rest, PSV 0 cmH2O and PEEP 0 cmH2O trial for 15 min.
  Interventions: Procedure: T-piece; Procedure: PSV 7 and PEEP 0; Procedure: PSV 0 and PEEP 0
- T-piece and PSV 0 PEEP 0 and PSV 7 PEEP 0 (Experimental): First T-piece trial for 15 min. After 10 min of rest, PSV 0 cmH2O and PEEP 0 cmH2O trial for 15 min. After 10 min of rest, PSV 7 cmH2O and PEEP 0 cmH2O trial for 15 min.
  Interventions: Procedure: T-piece; Procedure: PSV 7 and PEEP 0; Procedure: PSV 0 and PEEP 0
- PSV 0 PEEP 0 and PSV 7 PEEP 0 and T-piece (Experimental): First PSV 0 cmH2O and PEEP 0 cmH2O trial for 15 min. After 10 min of rest, PSV 7 cmH2O and PEEP 0 cmH2O trial for 15 min. After 10 min of rest, T-piece trial for 15 min.
  Interventions: Procedure: T-piece; Procedure: PSV 7 and PEEP 0; Procedure: PSV 0 and PEEP 0
- PSV 0 PEEP 0 and T-piece and PSV 7 PEEP 0 (Experimental): First PSV 0 cmH2O and PEEP 0 cmH2O trial for 15 min. After 10 min of rest, T-piece trial for 15 min. After 10 min of rest, PSV 7 cmH2O and PEEP 0 cmH2O trial for 15 min.
  Interventions: Procedure: T-piece; Procedure: PSV 7 and PEEP 0; Procedure: PSV 0 and PEEP 0
- PSV 7 PEEP 0 and T-piece and PSV 0 PEEP 0 (Experimental): First PSV 7 cmH2O and PEEP 0 cmH2O trial for 15 min. After 10 min of rest, T-piece trial for 15 min. After 10 min of rest, PSV 0 cmH2O and PEEP 0 cmH2O trial for 15 min.
  Interventions: Procedure: T-piece; Procedure: PSV 7 and PEEP 0; Procedure: PSV 0 and PEEP 0
- PSV 7 PEEP 0 and PSV 0 PEEP 0 and T-piece (Experimental): First PSV 7 cmH2O and PEEP 0 cmH2O trial for 15 min. After 10 min of rest, PSV 0 cmH2O and PEEP 0 cmH2O trial for 15 min. After 10 min of rest, T-piece trial for 15 min.
  Interventions: Procedure: T-piece; Procedure: PSV 7 and PEEP 0; Procedure: PSV 0 and PEEP 0

INTERVENTIONS:
Procedure: T-piece — Spontaneous breath trial with a T-piece
Procedure: PSV 7 and PEEP 0 — Spontaneous breath trial with a pressure support ventilation of 7 cmH2O and no positive end expiratory pressure
Procedure: PSV 0 and PEEP 0 — Spontaneous breath trial without pressure support ventilation and positive end expiratory pressure, with a patient intubated and connected to the ventilator

SUMMARY:
Assessment and comparison of three spontaneous breathing trials in five specific profiles of intensive care unit and perioperative patients. A physiological cross over study

DETAILED DESCRIPTION:
Mechanical ventilation is the most used organ replacement therapy in intensive care unit (ICU). After resolution of acute illness, separating the ventilator from the patient may be specially challenging. Before extubation, it is recommended to perform a spontaneous breathing trial (SBT) to evaluate the ability to sustain breathing with minimal or no support.

The way to carry out this step of the weaning process present important variation across regions of the world. Two techniques are preferentially used : the T-piece trial (oxygen supply without positive pressure) and low pressure support ventilation (PSV) from 6 to 10 cmH2O according to the airway humidification device.

The best strategy for successful weaning remains unknown, especially about specific subgroups of respiratory and neurological diseases.

Our aim is to assess which spontaneous breathing trial would best reproduce post-extubation inspiratory effort. We compare T-piece trial, PSV 7 cmH2O without positive end expiratory pressure (PEEP) and PSV 0 cmH2O without PEEP. Five specific profiles are evaluated : chronic obstructive pulmonary disease (COPD), severe brain injury, blunt thoracic trauma, post abdominal surgery and miscellaneous.

The hypothesis is that T-piece trial and PSV 0 CPAP 0 trial are the best for mimic inspiratory effort after extubation. However, we could highlight various results according to different subgroups of ICU patients. The final aim is to determine a personalized wean trial for each.

ELIGIBILITY:
Inclusion Criteria:

* ICU patient with invasive mechanical ventilation for at least 24 hours
* Physician decision to extubate and all criteria for ventilatory weaning must be present
* Resolution of disease acute phase for which the patient was intubated
* Conscious patient (Richmond Agitation-Sedation Scale (RASS) > 0), no sedation
* Good coughing effort, good swallowing, positive leak test (> 12% of tidal volume (VT))
* No important secretions
* No respiratory acidosis, adequate oxygenation (PaO2 / FiO2 > 150 mmHg and CPAP ≤ 8)
* Adequate pulmonary function (respiratory rate (RR) ≤ 35, negative inspiratory force (NIF) > 20 cmH2O, RR/VT < 105)
* Stable cardiovascular status (heart rate (HR) < 140 bpm, systolic blood pressure > 90 mmHg, no or minimal vasopressors)
* If severe brain injury, the VISAGE score must be ≥ 3 (visual pursuit, good swallowing, GCS > 10)

Exclusion Criteria:

* Obese patients with BMI ≥ 35 kg/m2
* Contraindication for nasogastric tube or esophageal manometric balloon placement
* Refusal of study participation or to pursue the study by the patient, no consent
* Pregnancy or breastfeeding
* Absence of coverage by the French statutory healthcare insurance system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Esophageal Pressure Time Product per minute (PTPes.min) | Day one
  In cmH2O.s/min. Assessment of patient's inspiratory effort. Integration of esophageal swing pressure over time, performed with a second-generation balloon esophageal catheter, immediately before and after each spontaneous breathing trial, before and 20 min after extubation

SECONDARY OUTCOMES:
Esophageal Pressure Time Product per minute (PTPes.min) | Day two
  In cmH2O.s/min. If esophageal catheter still in place, patient's inspiratory effort 24 hours after extubation
Esophageal Pressure Time Product per minute (PTPes.min) | Day three
  In cmH2O.s/min. If esophageal catheter still in place, patient's inspiratory effort 48 hours after extubation.

OTHER OUTCOMES:
Tidal impedance variation (TIV) assessed with Electrical Impedance Tomography | Day one
  In unit of impedance change (AU). Assessment of pulmonary volumes, only for the patients included in the center of Saint Eloi University hospital (ancillary study), immediately before and after each spontaneous breathing trial, before and 20 min after extubation.
End Expiratory Lung Impedance (EELZ) assessed with Electrical Impedance Tomography | Day one
  In unit of impedance change (AU). Assessment of pulmonary volumes, only for the patients included in the center of Saint Eloi University hospital (ancillary study), immediately before and after each spontaneous breathing trial, before and 20 min after extubation.
Global inhomogeneity index (GI) assessed with Electrical Impedance Tomography | Day one
  In percentage. Assessment of pulmonary volumes, only for the patients included in the center of Saint Eloi University hospital (ancillary study), immediately before and after each spontaneous breathing trial, before and 20 min after extubation.
Regional Ventilation Delay (RVD) index assessed with Electrical Impedance Tomography | Day one
  Assessment of pulmonary volumes, only for the patients included in the center of Saint Eloi University hospital (ancillary study), immediately before and after each spontaneous breathing trial, before and 20 min after extubation.
Subjective discomfort assessment with Numeric discomfort scale | Day one
  Visual numeric scale from 0 (no discomfort) to 10 (worst discomfort experienced), before and after each spontaneous breathing trial
Objective discomfort assessment with respiratory rate > 30 per min | Day one
  Before and after each spontaneous breathing trial
Post extubation respiratory management | Day three
  Physiotherapy (yes or no), oxygen therapy (yes or no, parameters), noninvasive ventilation (yes or no, parameters), the day of extubation, at 24h and 48h post extubation
Extubation success or failure | Day three
  Extubation success (no reintubation) or failure (reintubation) within 48h after extubation.

CONTACTS AND LOCATIONS:
Overall Officials: Samir Jaber, MD, PHD, Study Director — Montpellier University Hospital
Locations (1):
- Centre Hospitalier Universitaire Saint Eloi, Montpellier, Herault, France

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data will be made available upon a reasonable request
Supporting Information: Study Protocol
Time Frame: 12 months after the main publication
Access Criteria: Data are provided to qualified investigators free of charge. Required documents to request data include a summary of the research plan, request form, and institutional review board (IRB) review. Dataset will be shared after careful examination by the study board of investigators.

REFERENCES:
- [Background] Mahul M, Jung B, Galia F, Molinari N, de Jong A, Coisel Y, Vaschetto R, Matecki S, Chanques G, Brochard L, Jaber S. Spontaneous breathing trial and post-extubation work of breathing in morbidly obese critically ill patients. Crit Care. 2016 Oct 27;20(1):346. doi: 10.1186/s13054-016-1457-4. PMID 27784322
- [Derived] Capdevila M, De Jong A, Aarab Y, Vonarb A, Carr J, Molinari N, Capdevila X, Brochard L, Jaber S. Which spontaneous breathing trial to predict effort to breathe after extubation according to five critical illnesses: the cross-over GLOBAL WEAN study protocol. BMJ Open. 2023 Jul 12;13(7):e070931. doi: 10.1136/bmjopen-2022-070931. PMID 37438068